CLINICAL TRIAL: NCT01553110
Title: An Observational Study to Evaluate The Relationship of Nasal Mucus Properties and Symptoms in Acute Rhinosinusitis.
Brief Title: An Observational Study to Evaluate The Relationship of Nasal Mucus Properties and Symptoms
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM14200
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Acute Rhinosinusitis; Allergic Rhinitis
Keywords: Cold; Acute Rhinosinusitis; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Common Cold

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal Secretions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cold Population: Male and female subjects 12 years of age and older with acute nasal discharge fewer then 7 days. Patients must be symptomatic at screening.
- Allergic Rhinitis: Male and female subjects of 12 years of age and older with a history suggesting nasal allergic symptoms for at least 1 year. Patients must be symptomatic at screening.

SUMMARY:
This is a study to learn more about the common cold from studying the nasal secretions produced during a cold or episode of allergic rhinitis.

DETAILED DESCRIPTION:
This study involves collecting and analyzing nasal mucus to see if there are changes in mucus properties during the course of a cold or episode of allergic rhinitis. Outcome measures include SNOT20 questionnaire, nasal secretion collection, acoustic rhinometry on the fifth and fourteenth day of symptoms. The investigators will also collect SNOT20 questionnaires on the tenth and twenty-eighth day.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 12 years of age and older with acute nasal discharge fewer than 7 days or a history suggesting nasal allergic symptoms for at least 1 year. Internet access required during the course of the study. Patients must be symptomatic at screening.

Exclusion Criteria:

* Symptoms suggesting bacterial rhinosinusitis such as fever ≥ 101ºF/38.3ºC, facial swelling, and serve tooth pain. History of CRS or sinus/nasal surgery for this condition within 6 months before screening. History of respiratory signs and symptoms due to allergic rhinitis. Therapy with bronchodilators, nasal steroids, oral corticosteroids in the past 30 days. Therapy with antihistamines, nasal (Neti) washings, or decongestants in the past 24 hours. Use of any OTC cold or allergy medication 24 hours before study visits requires a 24 hour washout phase

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinics and Community
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-03; Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Nasal Secretion Collection | 10 minutes
  To measure the biophysical properties of nasal secretions for improved mucus clearance.

SECONDARY OUTCOMES:
Subjective nasal scoring | 10 Minutes
  The Sinus and Nasal Quality of Life Survey (SN-20) questionnaire assess the impact of infection on nasal symptoms, emotion, and activity on a scale of worsening symptoms scored 1 through 7 to provide a quantifiable score capable of comparing both disease severity and the impact of interventions on subjective complaints.
Nasal Volume | 15 Minutes
  Acoustic rhinometry is used to measure cross-sectional volume of the nasal cavity allowing the calculation of nasal volume.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce K Rubin, MEngr, MD, MBA, FRCPC, Principal Investigator — Virginia Commonwealth University School of Medicine; Melissa A Yopp, M.S.H.A, Study Director — Virginia Commonwealth University School of Medicine
Locations (1):
- Virginia Commonwealth University School of Medicine, Richmond, Virginia, United States